CLINICAL TRIAL: NCT00826371
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Ranibizumab (0.5 mg) in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration Over 12 Months
Brief Title: Evaluation of Safety and Efficacy of Once Monthly Ranibizumab Injections in Chinese Patients With Wet Age Related Macular Degeneration (AMD) Patients
Acronym: EXTEND II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002A2203
Record Dates: First submitted 2009-01-16; First posted 2009-01-22 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; Ranibizumab
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ranibizumab 0.5 mg

INTERVENTIONS:
Drug: ranibizumab 0.5 mg

SUMMARY:
The purpose of the study is to provide efficacy and safety data for monthly ranibizumab 0.5 mg intravitreal injections in Chinese patients with subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD). The study results will support the regulatory submission in China to make ranibizumab available for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese patients 50 years of age or greater.
* Patients with primary or recurrent subfoveal CNV secondary to AMD.
* Patients who have a BCVA score from 73 to 24 characters in the study eye.

Exclusion Criteria:

* Active, or history of, ocular inflammation or infection in the study eye within the last 30 days.
* Uncontrolled glaucoma in the study eye.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy of ranibizumab 0.5 mg by mean change in best-corrected visual acuity (BCVA) from Baseline to Month 4 as assessed with early treatment of diabetic retinopathy study (ETDRS) like charts at a distance of 4 meters. | 12 months

SECONDARY OUTCOMES:
To evaluate the effects of ranibizumab 0.5 mg on the change in BCVA from Baseline to Month 12. | 12 Months
To evaluate effects of ranibizumab 0.5 mg on retinal structure at Month 4 and Month 12 as assessed by fundus photography, fluorescein angiography, and optical coherence tomography. | 12 Months
To evaluate safety of ranibizumab 0.5 mg by rates of adverse events/SAEs, ophthalmic exams, tonometry, and changes in laboratory values/vital signs at Months 4 and 12. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- China (4):
  - Novartis Investigative Site, Beijing
  - Novartis Investigational Site, Chengdu
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai

REFERENCES:
- [Result] Zhao J, Li X, Tang S, Xu G, Xu X, Zhang F, Zhang M, Shamsazar J, Pilz S, Nieweg A. EXTEND II: an open-label phase III multicentre study to evaluate efficacy and safety of ranibizumab in Chinese patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration. BioDrugs. 2014 Dec;28(6):527-36. doi: 10.1007/s40259-014-0106-1. PMID 25012926